CLINICAL TRIAL: NCT03338335
Title: Ethnic Differences in Ischemia/Bleeding Risk Tradeoff During Antiplatelet Therapy After Drug-eluting Stent Implantation
Brief Title: Ethnic Differences and the Ischemia/Bleeding Risk of DAPT Duration
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hyo-Soo Kim, Professor, Seoul National University Hospital
Other Study IDs: DAPT
Record Dates: First submitted 2017-11-07; First posted 2017-11-09 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Coronary Artery Disease; Percutaneous Coronary Intervention; Dual Antiplatelet Therapy
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: prolonged DAPT — Dual antiplatelet therapy will be prescribed for more than 12 months

SUMMARY:
this study is an individual patient level meta-analysis of randomized clinical trials, to evaluate the influence of ethnicity, to study whether the relative tradeoff between ischemia and bleeding is distinct by ethnicity.

ELIGIBILITY:
Inclusion Criteria:

* patients enrolled in previous RCTs related to the duration of dural antiplatelet agent therapy

Ages: 19 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: individual participant data (IPD) meta-analysis of randomized controlled trials designed to investigate the efficacy and safety of shorter duration of DAPT with a longer duration DAPT in patients with ischemic heart diseases.
Sampling Method: Non-Probability Sample
Enrollment: 16000 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-03-31 (Estimated); Study Completion 2018-10-31 (Estimated)

PRIMARY OUTCOMES:
primary ischemic endpoint | 2 years
  major adverse cardiac events (MACE) defined as the composite of cardiac death, myocardial infarction, or definite/probable stent thrombosis
primary bleeding endpoints | 2 years
  major bleeding events

SECONDARY OUTCOMES:
all-cause death | 2 years
cardiac death | 2 years
non-cardiac death | 2 years
any myocardial infarction | 2 years
any stroke | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
This will be decided after the present analysis is completed.

REFERENCES:
- [Derived] Kang J, Park KW, Palmerini T, Stone GW, Lee MS, Colombo A, Chieffo A, Feres F, Abizaid A, Bhatt DL, Valgimigli M, Hong MK, Jang Y, Gilard M, Morice MC, Park DW, Park SJ, Jeong YH, Park J, Koo BK, Kim HS. Racial Differences in Ischaemia/Bleeding Risk Trade-Off during Anti-Platelet Therapy: Individual Patient Level Landmark Meta-Analysis from Seven RCTs. Thromb Haemost. 2019 Jan;119(1):149-162. doi: 10.1055/s-0038-1676545. Epub 2018 Dec 31. PMID 30597509